CLINICAL TRIAL: NCT06732531
Title: A Phase I/II, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of BH011 in Subjects With Recurrent High-Risk Non-Muscle-Invasive Bladder Cancer After Bacillus Calmette-Guérin
Brief Title: Safety, Tolerability, and Preliminary Efficacy of BH011 in Subjects With Non-Muscle-Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhuhai Beihai Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH011-I/II-1001; CTR20220208 (Other: CENTER FOR DRUG EVALUATION, NMPA)
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer; Non Muscle Invasive
Keywords: BH011; High-Risk Non-Muscle-Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BH011 (Experimental): BH011 is administered intravesically through a urinary catheter and is retained in the bladder for 1 hour.
  Interventions: Drug: BH011

INTERVENTIONS:
Drug: BH011 — BH011 is administered intravesically through a urinary catheter and is retained in the bladder for 1 hour. It was administered once a week for 6 weeks during the induction treatment period and once a month for 12 months during the maintenance treatment period.
  Other Names: Docetaxel

SUMMARY:
The purpose of this study is to determine the safety and tolerability of intravesical BH011 in patients with high-risk non-muscle invasive bladder cancer（NMIBC） after Bacillus Calmette-Guerin（BCG） failure and to assess the preliminary efficacy.

DETAILED DESCRIPTION:
The plan is to study the safety and preliminary efficacy of BH011 in High-Risk NMIBC patients who failed BCG therapy. Most patients with NMIBC is (Cis, Cis with Ta and/or T1, high grade Ta or T1 with frequent or uncontrolled recurrences) who have failed BCG intravesical therapy (standard of care) usually have no other choice but to proceed to cystectomy. Cystectomy is a surgery associated with major morbidity, mortality and quality of life issues. Morbidity and long term tedious medical care will be for the rest of the patient's life span. Most patients at this stage do not show signs of disease progression into the muscle layer or of metastasis, making surgery a very difficult decision. BH011 will serve to provide a therapeutic alternative for this patient population in need.

In this study, patients will begin treatment with BH011 2-8 weeks after TURBT and will be administered once weekly for 6 weeks during the induction treatment period and once monthly for 12 months in the maintenance treatment period. Patients will undergo cystoscopy, urine cytology, and biopsy every 3 months for up to 24 months to confirm clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were fully informed about the study and voluntarily signed an informed consent form and were willing to complete the trial in accordance with the protocol process.
2. Male or female, ≥18 years of age at time of informed consent.
3. First TURBT completed within 12 weeks prior to the first dose, histologically confirmed diagnosis of non-muscle invasive bladder cancer and classified as high risk according to the European Association of Urology 2020 version of the Non-Muscle Invasive Bladder Cancer Guidelines.
4. Patients who had failed intravesical administration of BCG prior to enrolment and were not candidates for or refused radical cystectomy.BCG failures included BCG refractory, recurrence after BCG, BCG non-responsive, and BCG intolerant;
5. After TURBT, it is confirmed that the tumour has been completely removed from the bladder. A second TURBT is required for the following: confirmed or suspected incomplete resection of the tumour by TURBT; absence of muscularis propria tissue in the first resection of the tumour specimen, except for TaLG/G1 tumours or primary carcinoma in situ; and stage T1 bladder tumours. A second TURBT is recommended 2 to 6 weeks after the initial TURBT.
6. Eastern Cooperative Oncology Group (ECOG) score 0 to 1.
7. Expected survival ≥ 6 months.
8. The major organs are functioning well, i.e. the following criteria are met:

   * Bone marrow function: hemoglobin (HGB) ≥80 g/L, platelet count (PLT) ≥100×109/L, absolute neutrophil count (ANC) ≥1.5×109/L.
   * Liver function: serum total bilirubin ≤ 1.25 x upper limit of normal (ULN) (or 2.5 × ULN in case of constitutional hepatic dysfunction jaundice [Gilbert's syndrome]), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN.
   * Renal function: creatinine clearance ≥30 mL/min (Cockcroft-Gault formula) or serum creatinine ≤2.0 mg/dL.

Exclusion Criteria:

1. Patients with muscle-invasive bladder cancer (T2-T4).
2. Patients with urothelial carcinoma of the upper or lower urinary tract, and/or lymph node metastases.
3. Patients with a history of vesicoureteral reflux.
4. Patients with other malignancies within 2 years, except locally curable (cured) cancers, e.g. basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix.
5. Patients who have not recovered (toxicity assessment remains > Grade 1 or has not recovered to baseline levels) from toxic reactions (other than malaise, alopecia) associated with prior antineoplastic therapy; patients who have not recovered to Grade 0-1 (CTCAE 5.0) within 3 days prior to the first dose for the following: uncontrolled acute and chronic infections, e.g., pneumonitis, biliary tract infections, hepatitis B virus infections, and hepatitis C virus infections; Respiratory distress; acute and chronic kidney injury; nephrotic syndrome; bladder perforation; urinary tract obstruction.
6. Patients with severe or uncontrolled cardiac disease requiring treatment, including: a) severe arrhythmias (ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block, etc.); b) history of myocardial infarction, unstable angina pectoris, angioplasty, or coronary artery bridging surgery within 6 months prior to the first dose of the study drug; c) New York Heart Association (NYHA) class III or IV congestive heart failure (see Appendix 4); d) 12-lead electrocardiography: corrected QTc intervals: QTc > 450 ms in men and QTc > 470 ms in women (QTc intervals were calculated using the Fridericia formula).
7. Patients with uncontrolled hypertension on treatment (defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg).
8. Patients with peripheral neuropathy > grade 1.
9. Patients with known or suspected hypersensitivity to docetaxel, its excipients or similar drugs.
10. Patients previously treated with docetaxel.
11. Patients with previous extensive radiotherapy to the pelvis (radiotherapy > 30% of the bone marrow area).
12. Patients who have undergone major surgical treatment within 28 days prior to the first dose, or who have failed to recover to ≤ grade 2 from adverse effects of any such procedure.
13. Patients who have received intravesical therapy within 28 days prior to the first dose (immediate chemotherapy infusion after previous and current electrodes is permitted).
14. Patients receiving antitumor therapy such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, biologic therapy, and herbal medicine within 28 days or 5 half-lives of the drug, whichever is longer, prior to the first dose.
15. Patients who have participated in any other clinical interventional trial treatment (other than patients enrolled in a study with overall survival follow-up) within 28 days or 5 half-lives, whichever is longer, prior to the first dose.
16. Patients who plan to receive other anticancer treatments or other investigational drugs during the study period.
17. Pregnant or breastfeeding female patients. Positive blood pregnancy test in females of childbearing potential within 7 days prior to first dose; Any male and female patient of childbearing potential refuses to use a contraceptive method with an annual failure rate of <1% (contraceptive methods with an annual failure rate of <1% include bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives that suppress ovulation, hormone-releasing intrauterine devices (IUDs), and copper-containing IUDs, or condoms) throughout the duration of the trial and for a period of 30 days after the last study dose. In the judgment of the investigators, a patient is defined as having the ability to procreate as he/she is biologically capable of having children as well as having a normal sex life. Female patients who are not of childbearing potential (i.e., meet at least 1 of the following criteria):

    * Has had a hysterectomy or bilateral oophorectomy, or
    * Medically diagnosed with ovarian failure, or
    * Medically diagnosed as post-menopausal (menopause for at least 12 consecutive months in the absence of pathologic or physiologic causes).
18. Patients with known history of psychiatric disorders, substance abuse, drug and alcohol addiction, and impairments in adherence.
19. Any other patients who, in the opinion of the investigator, would result in unnecessary risk to the subject and are therefore unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From first dose to 30 days after last dose
  Adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
3 month Complete Response Rate (CRR) | 3 months
  Complete Response rate is defined as the percentage of participants achieving a CR at 3 months post-treatment. It will be measured by determining the percentage of participants without presence of high-grade disease using results from cystoscopy and urine cytology at any time point.

SECONDARY OUTCOMES:
6 month Complete Response Rate (CRR) | 6 months
  Complete Response rate is defined as the percentage of participants achieving a CR at 6 months post-treatment. It will be measured by determining the percentage of participants without presence of high-grade disease using results from cystoscopy and urine cytology at any time point.
Recurrence-Free Survival (RFS) | up to 24 months
  RFS is defined as the time from the first study treatment to the presentation of the first pathologically confirmed high-risk non-muscle invasive bladder cancer (T1, CIS, or high-grade Ta) recurrence or death from any cause, whichever occurred earliest.
Progression-Free Survival (PFS) | up to 24 months
  PFS is defined as the time from the first study treatment to the occurrence of the first bladder cancer infiltration into the muscularis propria, lymphatic metastasis, distant metastasis, or death from any cause, whichever occurred earliest.
Recurrence-Free Survival Rate | up to 24 months
  The RFS rate is defined as the rate of subjects without pathologically confirmed high-risk non-muscle invasive bladder cancer (T1, CIS, or high-grade Ta) recurrence or death from any cause.
Progression-Free Survival Rate | up to 24 months
  The PFS rate is defined as the rate of subjects free of bladder cancer infiltration into the muscularis propria, lymphatic metastasis, distant metastasis, or death from any cause.
Pharmacokinetic of BH011 | Weeks 1 and 6 of dosing
  Maximum Concentration (Cmax)
Pharmacokinetic of BH011 | Weeks 1 and 6 of dosing
  Time to Cmax (Tmax)
Pharmacokinetic of BH011 | Weeks 1 and 6 of dosing
  Area Under the Curve From Time 0 Hours to Last Quantifiable Concentration (AUC0-last)
Pharmacokinetic of BH011 | Weeks 1 and 6 of dosing
  Area Under the Curve From Time 0 Hours to Infinity (AUC0-inf)
Pharmacokinetic of BH011 | Weeks 1 and 6 of dosing
  Apparent Terminal Elimination Half-Life (t1/2)
Pharmacokinetic of BH011 | Weeks 1 and 6 of dosing
  Apparent Total Clearance (CL)
Pharmacokinetic of BH011 | Weeks 1 and 6 of dosing
  Apparent Volume of Distribution (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wei, Study Director — Zhuhai Beihai Biotech Co., Ltd
Locations (6):
- China (6):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality